CLINICAL TRIAL: NCT00108056
Title: A Phase I Trial of Enzastaurin (LY317615) in Patients With Recurrent Gliomas
Brief Title: Enzastaurin to Treat Recurrent Brain Tumor
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 050136; 05-C-0136; NCT00112788 (obsolete NCT alias)
Record Dates: First submitted 2005-04-12; First posted 2005-04-13 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2014-04-01

CONDITIONS: Glioma
Keywords: Brain; Tumor; Malignant; Therapy; Progression; Malignant Brain Tumor; Malignant Glioma; Glioma
MeSH Terms: conditions — Glioma; Neoplasms; Disease Progression; Brain Neoplasms | interventions — enzastaurin

INTERVENTIONS:
Drug: Enzastaurin (LY317615) monohydronchloride

SUMMARY:
This study will examine the safety of a twice-a-day dosing regimen of the experimental drug Enzastaurin in patients with malignant glioma (a cancerous brain tumor) who are and who are not taking certain anti-seizure medicines. Enzastaurin may prevent the formation of new blood vessels that tumors need to grow. It has shown some effect against brain tumors in animals and in some patients with recurrent gliomas. This study will see if the drug can help patients with gliomas and how much drug they should be given.

Patients 18 years of age and older with malignant glioma that has recurred after standard therapy may be eligible for this study. Candidates are screened with a physical examination, blood and urine tests, magnetic resonance imaging (MRI) or computed tomography (CT) scans, and an electrocardiogram.

Participants are divided into two groups of patients-those who are and those who are not taking certain anti-seizure medications-in order to determine if the anti-seizure medication alters the way the body handles Enzastaurin. Patients in both groups are further divided into different dosing regimens: some in each group take Enzastaurin once a day for 3 weeks, followed by twice a day for 3 weeks; others in the group take the drug twice a day for 3 weeks followed by once a day for 3 weeks. The medication is taken by mouth every day. Treatment is given in 6-week cycles and may continue for 1 year unless the tumor grows or the patient develops unacceptable drug side effects. In addition to drug treatment, patients have the following tests and procedures:

* Medical history, physical, and neurological examinations every 3 weeks during the first cycle and then every 6 weeks.
* MRI or CT scan of the head before starting each new cycle. MRI uses a magnetic field and radio waves to produce images of body tissues and organs. CT uses x-rays to provide 3-dimensional views of the part of the body being studied. For both procedures, the patient lies on a table that slides into the cylindrical scanner.
* Routine blood tests every week during the first cycle and every 3 weeks after that.
* Electrocardiogram on days 21 and 42 of the first cycle, just before taking the drug and 30 minutes and 4 hours after taking the drug.
* Pharmacokinetic studies within 3 days of day 21 of the first cycle. Several blood samples are drawn to measure levels of Enzastaurin. Patients taking the drug once a day have blood samples drawn before the morning dose and 1, 2, 4, 6 and 24 hours after the dose. Patients taking the drug twice a day have samples drawn before the morning dose, at 1, 2, 4, 6 and 12 hours after the dose, and then 12 hours after the evening dose. In addition, on day 1 an extra tube of blood is drawn at the time of the Enzastaurin dose and 4 hours later.
* Dynamic MRI with spectroscopy or PET. These tests are done to help distinguish live tumor from dying tumor. The experience of dynamic MRI with spectroscopy is the same as standard MRI and is done at the same time as the standard procedure. PET uses a radioactive substance to show cellular activity in specific tissues of the body. The patient is given an injection of a sugar solution in which a radioactive isotope has been attached to the sugar molecule. A special camera detects the radiation emitted by the radioisotope, and the resulting images show how much glucose is being used in various parts of the body. Because rapidly growing cells, such as tumors, take up and use more glucose than normal cells do, this test can be used to show active tumors.

DETAILED DESCRIPTION:
BACKGROUND:

Enzastaurin is a macrocyclic bisindolylmaleimide which disrupts the intrinsic phosphotransferase activity of conventional and novel PKC isoforms via an interaction at the ATP binding site, displays selectivity in inhibiting the isoforms.

Preclinical studies demonstrate potent anti-angiogenic activity of enzastaurin and studies in normal volunteers and solid tumor patients demonstrate the drug is very well tolerated at doses that achieve a biologically active serum concentration.

OBJECTIVES:

To establish the maximally tolerated dose of enzastaurin in patients with refractory primary brain tumors not on any enzyme-inducing anti-epileptic drugs (EIAED) and for patients on EIAEDs.

To determine if twice a day dosing results in higher systemic exposure of enzastaurin and its metabolites than once a day dosing in patients not on EIAEDs and those on EIAEDs.

To obtain exploratory data regarding the relationship between the activity of the PKC-b pathway (specifically GSK3-b activation) in peripheral blood mononuclear cells of treated patients and clinical outcome.

To obtain exploratory information about the anti-tumor activity of enzastaurin at the higher doses specified in this protocol.

ELIGIBILITY:

Patients with histologically proven malignant glioma will be eligible for this protocol.

DESIGN:

Patients will be stratified into Group A or Group B based on their concomitant medications. Patients who are on enzyme inducing anti-epileptic drugs such as phenytoin, carbamazepine or trileptal will be enrolled into Group B while patients who meet the eligibility criteria and are not on any enzyme inducers, will be entered into Group A.

As of December 2005, three DLT's were observed at dose level 1 and it was determined that this was not a tolerable dose. A third dose level has been added using a lower dose for Group A patients only. Twelve patients will be entered at the third dose level in Group A only.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with histologically proven malignant glioma will be eligible for this protocol. Malignant glioma include glioblastoma multiforme (GBM), anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), or malignant glioma NOS (not otherwise specified). Additionally, patients with primitive neuroectodermal tumors (PNETs) of the central nervous system, progressive low-grade gliomas and radiographically diagnosed brain stem gliomas refractory to standard treatment will be eligible.

Patients must have unequivocal evidence for tumor progression by MRI or CT scan. This scan should be performed within 14 days prior to registration and on a steroid dosage that has been stable for at least 5 days. If the steroid dose is increased between the date of imaging and registration a new baseline MR/CT is required. The same type of scan, i.e., MRI or CT must be used throughout the period of protocol treatment for tumor measurement.

Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:

1. <TAB>They have recovered from the effects of surgery.
2. <TAB>Residual disease following resection of recurrent tumor is not mandated for eligibility into the study. To best assess the extent of residual disease post-operatively, a CT/ MRI should be done:

   * no later than 96 hours in the immediate post-operative period or
   * at least 4 weeks post-operatively, and
   * within 14 days of registration, and
   * on a steroid dosage that has been stable for at least 5 days.

   If the 96 hour scan is more than 14 days before registration, the scan needs to be repeated. If the steroid dose is increased between the date of imaging and registration, a new baseline MRI/CT is required on a stable steroid dosage for at least 5 days.

   Patients must have failed prior radiation therapy and must have an interval of greater than or equal to 4 weeks from the completion of radiation therapy to study entry.

   All patients must sign an informed consent indicating that they are aware of the investigational nature of this study.

   Patients must be greater than or equal to 18 years old, and with a life expectancy greater than 8 weeks.

   Patients must have a Karnofsky performance status of greater than or equal to 60.

   Patients must have recovered from the toxic effects of prior therapy: 2 weeks from any noncytotoxic investigational agent, 4 weeks from prior cytotoxic therapy, two weeks from vincristine, 6 weeks from nitrosoureas, 3 weeks from procarbazine administration, and 1 week for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count). Any questions related to the definition of non-cytotoxic agents should be directed to the Study Chair.

   Patients must have adequate bone marrow function (WBC greater than or equal to 3,000/micro l, ANC greater than or equal to 1,500/mm(3), platelet count of greater than or equal to 100,000/mm(3), and hemoglobin greater than or equal to10 gm/dl), adequate liver function (SGOT and bilirubin less than or equal to 2 times ULN), and adequate renal function (creatinine less than or equal to 1.5 mg/dL and/or creatinine clearance greater than or equal to 60 cc/min) before starting therapy. These tests must be performed within 14 days prior to registration. Eligibility level for hemoglobin may be reached by transfusion.

   Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patients' ability to tolerate this therapy

   This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender. No exclusion to this study will be based on race. Minorities will actively be recruited to participate.

   Patients must practice adequate contraception.

   Prior treatment with an enzyme inducing antiepileptic drug must have been discontinued at least 14 days prior to study entry for Group A patients.

   EXCLUSION CRITERIA:

   Patients who, in the view of the treating physician, have significant active cardiac, hepatic, or renal diseases are ineligible.

   No concurrent use of other standard chemotherapeutics or investigative agents.

   <TAB>

   Patients known to have an active malignancy (except non-melanoma skin cancer or carcinoma in-situ of the cervix).

   Patients who have an active infection requiring IV antibiotics.

   Patients who are pregnant or breast feeding.

   Patients who have any disease that will obscure toxicity or dangerously alter drug metabolism.

   QTc with Bazett's correction that is unmeasurable, or greater than or equal to 460 msec on screening ECG. If a patient has QTc greater than or equal to 460 msec on screening ECG, a second screen ECG may be repeated at least 24 hours apart. The average QTc from the 2 screening ECGs must be less than 460 msec in order for the patient to be eligible for the study.

   EKG demonstrating clincically significant arrythmia (multifocal premature ventricular contraction [PVC], bigeminy, trigeminy, ventricular tachycardia, bradycardia) that is symptomatic or requires treatment (CTCAE grade 3), or asymptomatic sustained ventricular tachycardia.

   Patients who have baseline EKGs suggestive of past or present cardiac ischemia will not be eligible unless they have an appropriate (as defined by the P.I. of this trial) negative cardiac work up (i.e. echocardiogram, stress test).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-04-07; Primary Completion 2014-04-01 (Actual); Study Completion 2014-04-01 (Actual)

PRIMARY OUTCOMES:
To establish the maximally tolerated dose of enzastaurin in patients with refractory primary brain tumors not on any enzyme-inducing anti-epileptic drugs (EIAED) and for patients on EIAEDs.

CONTACTS AND LOCATIONS:
Overall Officials: Teri N Kreisl, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barker D, Wright E, Nguyen K, Cannon L, Fain P, Goldgar D, Bishop DT, Carey J, Baty B, Kivlin J, et al. Gene for von Recklinghausen neurofibromatosis is in the pericentromeric region of chromosome 17. Science. 1987 May 29;236(4805):1100-2. doi: 10.1126/science.3107130.
- [Background] Bigner SH, Bjerkvig R, Laerum OD. DNA content and chromosomal composition of malignant human gliomas. Neurol Clin. 1985 Nov;3(4):769-84. PMID 3001489
- [Background] Moss AR. Occupational exposure and brain tumors. J Toxicol Environ Health. 1985;16(5):703-11. doi: 10.1080/15287398509530780. PMID 4093991